CLINICAL TRIAL: NCT00494650
Title: Cognitive Behavioral Treatment of Post-Traumatic Stress Disorder in Clients With Severe Mental Illness (in New Jersey)
Brief Title: Cognitive Behavioral Treatment for Post-Traumatic Stress Disorder in People With Additional Serious Mental Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH064662-02 (NIH); R01MH064662-02 (NIH); DSIR 83-ATIT
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive cognitive behavioral therapy.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- 2 (Active Comparator): Participants will receive brief PTSD treatment.
  Interventions: Behavioral: Brief PTSD treatment

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — CBT will include 12 to 16 counseling sessions, occurring weekly or every other week. Participants will learn about PTSD and ways to decrease anxiety associated with PTSD by completing homework assignments and practicing skills learned in counseling sessions.
  Arms: 1
Behavioral: Brief PTSD treatment — Brief PTSD treatment will include three weekly meetings with a therapist. Participants will learn about PTSD, how symptoms may be affecting their lives, and a technique for reducing anxiety associated with PTSD.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of tailored cognitive behavioral therapy in treating post-traumatic stress disorder in people with additional mental illnesses.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is an anxiety disorder that can develop after experiencing a terrifying event or ordeal in which grave physical harm occurred or was threatened. People with PTSD have persistent frightening thoughts and memories about the traumatic event and may experience sleep problems, feel detached or numb, or be easily startled. Studies have shown that PTSD occurs at high rates among people with serious mental illnesses (SMI), such as bipolar disorder, schizophrenia, and major depression. Research has also proven that cognitive behavioral therapy (CBT) is an effective PTSD treatment for caucasians living in rural areas when it is administered by a PhD-level clinician. It is not clear, however, how successful this treatment will be when it is delivered to a minority population by frontline mental health clinicians in an urban setting. This study will evaluate the effectiveness of tailored CBT in treating PTSD in people with additional mental illnesses who live in urban areas of New Jersey.

Participants in this 4- to 5-month open-label study will be randomly assigned to receive either brief PTSD treatment or CBT. Participants assigned to brief PTSD treatment will have three meetings with a therapist per week. Participants will learn about PTSD, how symptoms may be affecting their lives, and a technique for reducing anxiety associated with PTSD. Participants assigned to CBT will attend 12 to 16 counseling sessions per week or every other week. Participants will learn about PTSD and ways to decrease anxiety associated with PTSD by completing homework assignments and practicing skills learned in counseling sessions. Outcomes will be assessed for all participants through interviews that will occur immediately post-treatment, 6 months post-treatment, and 1 year post-treatment.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00053690

ELIGIBILITY:
Inclusion Criteria:

* Meets New Jersey definition of severe mental illness (SMI), which includes a DSM-IV diagnosis of an SMI; within the 3 to 6 months prior to study entry, functional limitations in major life activities that would be appropriate for the client's developmental stage; and within 2 years prior to study entry, two or more treatment episodes of greater intensity than outpatient services (such as inpatient, emergency, or partial hospitalization care, or a single episode lasting 3 months or more) OR a normal living situation disrupted to the point that supportive services were required to maintain the patient in their home or residence, or law enforcement officials were required to intervene
* DSM-IV Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depression (as determined by Structured Clinical Interview)
* Diagnosis of current severe PTSD at baseline assessment (as determined by a score greater than 65 on a Clinician Administered PTSD Scale)
* Speaks English

Exclusion Criteria:

* Current diagnosis of alcohol or drug dependence
* Hospitalization or suicide attempt in the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Knowledge of PTSD and effectiveness in correcting faulty, trauma-related beliefs | Measured post-treatment and at 6- and 12-month follow-ups
Depression, anxiety, and other psychiatric symptoms | Measured post-treatment and at 6- and 12-month follow-ups
PTSD diagnoses and symptom severity | Measured post-treatment and at 6- and 12-month follow-ups

SECONDARY OUTCOMES:
Total cost for mental health and substance abuse treatment services utilization within the University Behavioral Health Care system | Measured post-treatment and at 6- and 12-month follow-ups
Quality of life and community functioning | Measured post-treatment and at 6- and 12-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Kim T. Mueser, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (5):
- United States (5):
  - United Behavioral HealthCare (UBHC): Partial Hospital Program, Monmouth Junction, New Jersey
  - University Behavioral HealthCare (UBHC) Adult Outpatient Psychiatric Services, New Brunswick, New Jersey
  - University Behavioral HealthCare (UBHC) Extended Treatment, New Brunswick, New Jersey
  - University Behavioral HealthCare (UBHC) Extended Treatment Division - Adult Outpatient Psychiatric Services, Newark, New Jersey
  - University Behavioral HealthCare (UBHC) Extended Treatment Division - Partial Hospital Program, Newark, New Jersey

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Mueser KT, Gottlieb JD, Xie H, Lu W, Yanos PT, Rosenberg SD, Silverstein SM, Duva SM, Minsky S, Wolfe RS, McHugo GJ. Evaluation of cognitive restructuring for post-traumatic stress disorder in people with severe mental illness. Br J Psychiatry. 2015 Jun;206(6):501-8. doi: 10.1192/bjp.bp.114.147926. Epub 2015 Apr 9. PMID 25858178